CLINICAL TRIAL: NCT02311855
Title: Duration of Immune Response to Influenza Vaccination in Patients With Rheumatoid Arthritis Receiving Treatment With Biologic Agents
Brief Title: Duration of Immune Response to Influenza Vaccination in Patients With RA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Donald A Raddatz, Attending Physician, Department of Medicine - Rheumatology, Bassett Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1076
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Influenza vaccination (Other): all patients are vaccinated per protocol
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Each participant will have a blood draw to measure the antibody titres influenza strains covered by the 2014-2015 influenza vaccine at three different time points:
  Visit 1- Baseline/prior to vaccination Visit 2- 4-6 weeks post-vaccination Visit 3- end of influenza season (April-May)
  At Visit 1, after the baseline blood draw, all participants will be vaccinated by Research staff in order to standardize the time from Baseline blood draw to vaccination. Participants aged 65 and older will be offered the extra strength version of the vaccine, which is usual care. Participants under the age of 65 will be given the usual strength vaccine. All patients will be given the intramuscular (IM) vaccine.
  Other Names: Fluzone; Fluzone High Dose

SUMMARY:
The main objective is to evaluate the strength and duration of immune response after influenza vaccination in patients with Rheumatoid Arthritis (RA) receiving treatment with biological agents as compared to a group healthy controls who do not have RA. Influenza vaccine titers will be drawn 3 times: at Baseline(prior to vaccination), 4-6 weeks post vaccination, and 5-6 months post vaccination. Influenza vaccination will be done at the baseline visit after the baseline blood draw.

DETAILED DESCRIPTION:
Aims:

* Evaluate the strength and duration of immune response after influenza vaccination in patients with Rheumatoid Arthritis (RA) receiving treatment with biological agents.
* Evaluate for predictors of immune response such as age, gender, disease duration, type of the biological agent(s) used, duration of the treatment, and type of treatment in the past.
* Assess the efficacy of vaccine response in this population by recording proportion of patients who contracted influenza illness despite vaccination. The result of the study may provide more information regarding which situations inadequate immune response by strength or duration would most likely to be expected. This may help lay some groundwork for future studies looking at the use of booster vaccinations in this population

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (RA Patients)

* Patients with RA receiving treatment with an Anti-T Cell or Anti-TNF biological agent
* Age 40-75

Inclusion Criteria (Healthy Controls):

* Age 40-75

Exclusion Criteria:

Exclusion criteria (RA Patients)

* Known hypersensitivity/allergy influenza vaccine
* Chronic debilitating conditions (such as end-stage Chronic Obstructive Pulmonary Disease (COPD), Congestive Heart Failure (CHF), liver disease, Chronic Kidney Disease (CKD) )
* Active malignancy at time of vaccination
* Pregnancy and lactation
* Known HIV
* Active infection at time of vaccination
* Recent acute illness (within 1 month prior to vaccination)

Exclusion Criteria(Healthy Controls):

* Known autoimmune conditions
* Chronic use of immunosuppressant treatments
* Known hypersensitivity/allergy influenza vaccine
* Chronic debilitating conditions (such as end-stage COPD, CHF, liver disease, CKD)
* Active malignancy at time of vaccination
* Pregnancy and lactation
* Known HIV
* Active infection at time of vaccination
* Recent acute illness (within 1 month prior to vaccination)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Initial Immune response | 4-6 weeks post vaccination
  proportion of subjects with at least a 4-fold increase in titer at 4-6 weeks postvaccination to this year's influenza vaccine antigens;
Total proportion of seroconversion | 6 months post vaccination
  proportion of subjects with a persistent level of antibodies for influenza at the end of influenza period

SECONDARY OUTCOMES:
Occurrence of influenza infection | 6 months post vaccination
  proportion of patients who are diagnosed with confirmed influenza despite vaccination
Occurrence of flu-like illnesses | 6 months post vaccination
  proportion of patient who developed influenza-like symptoms (defined as two or more of the following: cough, myalgias, fever, arthralgias, throat pain, headache, nasal congestion).

CONTACTS AND LOCATIONS:
Overall Officials: Donald Raddatz, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No